CLINICAL TRIAL: NCT05806424
Title: Investigation of Awareness Levels of Women Living in Turkey About Kegel Exercises and Pelvic Floor Muscles
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Other Study IDs: Kegel Exercises Pelvic Floor
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Female Sexual Dysfunction
Keywords: exercise; kegel exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pelvic muscle awareness
- not pelvic muscle awareness

SUMMARY:
Pelvic floor disorders affect millions of women and their lives in our country and around the world. Along with many factors such as age, obesity, menopause, smoking, number of births and mode of delivery, there is an increase in the prevalence of pelvic floor disorders. Pelvic floor disorders (urinary/fecal incontinence, pelvic organ prolapse, chronic pelvic pain, sexual dysfunction) negatively affect women, their families, caregivers of individuals who cannot meet their own needs, and society in many ways. Treatment of pelvic floor disorders is very costly on a community basis. An effective process is carried out with the use of non-pharmacological traditional and complementary therapies instead of invasive or pharmacological treatment in the early period of the treatment of symptoms of pelvic floor disorders.

DETAILED DESCRIPTION:
Pelvic floor muscle training has a positive effect on voiding functions by strengthening the urogenital sphincter muscle. One of the commonly used methods for pelvic floor muscle training is the so-called Kegel exercise.

Sexual life, with its personal and social aspects, is an inseparable part of human beings in general, it is one of the most important factors in human life and happiness, especially in family life. Sexuality positively integrates and enriches the somatic, emotional, intellectual and social aspects of individuals, and develops personality, communication and love.

Kegel exercises; It is a method for strengthening the muscles that fix the bladder, intestines and genital organs in the pelvis and control their movements. These are tightening and relaxation exercises that strengthen the pelvic muscles. Like all voluntary muscles, the pelvic floor muscles are muscles that get stronger and develop as they work. Women of all ages need to have strong pelvic floor muscles.

ELIGIBILITY:
Inclusion Criteria:

* Living in Turkey
* Women aged 18 and over
* Having an active sex life

Exclusion Criteria:

* Having a disease affecting the pelvic floor muscles
* Having pelvic surgery in the last 6 months
* Being receiving sexual therapy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Kegel Exercises and Pelvic Floor Muscles
Study Population: Individuals who will participate in the study will be reached through online platforms. A questionnaire will be sent to the participants via the Google search engine and they will be asked to fill it out.
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2023-10-21 (Actual); Primary Completion 2023-10-21 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Demographic Information: | one day
  It was used to measure the general knowledge of the participants and their knowledge of knowing and applying Kegel exercises.
  Whether there is information about the pelvic floor muscles and Kegel exercises, the source of this information, whether the exercises are applied, which one is applied, the reason for the application, how long it is applied, whether the application is continued, from whom the training is received, how it is applied, whether it has positive effects. It is a questionable scale.
Female sexual function scale (FSFI) | one day
  The sexual functions of each subject included in the study were analyzed using the Female Sexual Function Index (FSFI). In the structure of the scale; There are 6 sub-dimensions: desire, arousal, lubrication (lubrication, wetting), orgasm, satisfaction and pain. Each item is scored from zero to 5. Accordingly, the highest raw score that can be obtained from the scale is 95.0 and the lowest raw score is 40. The reliability of the test was evaluated in two ways; Internal consistency and test-retest reliability were determined separately for 6 sub-dimensions with Cronbach's Alpha and their values were found to be 0.82 and higher.
Sexual Life Quality Scale- Female: | one day
  Each item is expected to be answered by considering the sexual life in the last four weeks. In scoring the scale, each question is scored between 1 and 6. The range of points that can be obtained from the scale is between 18 and 108. The scores of items 1, 5, 9, 13 and 18 must be reversed before the total score can be calculated. In order to convert the total scale score to 100 (raw score-18 from the scale), the formula x100/90 should be used. A high score from the scale indicates that the quality of sexual life is good.

SECONDARY OUTCOMES:
Beck Anxiety Scale | one day
  It is a self-report scale that determines the frequency of anxiety symptoms experienced by individuals. It is a Likert-type scale consisting of 21 items and scored between 0-3. The high scores obtained from the scale indicate the severity of the anxiety experienced by the individual. If the scores obtained from the scale are in the range of 0-7 points, it is considered as minimal anxiety / normal, between 8-15 points as mild anxiety, between 16-25 points as moderate anxiety, and between 26-63 points as severe anxiety. Although it is not certain, it is generally recommended to start medical treatment for individuals above 16 points. The treatment should be given by looking at the clinical condition of the patient as well as the score obtained from the scale.

CONTACTS AND LOCATIONS:
Locations (1):
- HAZAL genç, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Khosravi A, Riazi H, Simbar M, Montazeri A. Effectiveness of Kegel exercise and lubricant gel for improving sexual function in menopausal women: A randomized trial. Eur J Obstet Gynecol Reprod Biol. 2022 Jul;274:106-112. doi: 10.1016/j.ejogrb.2022.05.022. Epub 2022 May 21. PMID 35640438